CLINICAL TRIAL: NCT00559390
Title: Metabolic Syndrome in PCOS: Precursors and Interventions
Brief Title: Research Study for Children With a Mother or Sister With Polycystic Ovary Syndrome
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northwestern Memorial Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Andrea Dunaif, Principal Investigator, Northwestern University
Other Study IDs: 0956-023; R01DK040605 (NIH); DK73411
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Precursors to PCOS
Keywords: Polycystic Ovary Syndrome; Metabolic Syndrome; PCOS; children; girls; daughters; sisters; irregular periods
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Menstruation Disturbances

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Serum and Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-PCOS: First degree relatives, either sisters or daughters, of women with Polycystic Ovary Syndrome.
- Controls: Sisters and daughters of women who do not have PCOS

SUMMARY:
In this study, we want to find out more about polycystic ovary syndrome(PCOS). This is a common problem in about 7% of teenage girls. Problems may include irregular periods, extra hair on the face, chest and back areas. It seems that PCOS is related to a high level of male hormones and to another problem called metabolic syndrome(MBS). People with MBS may have high blood pressure, low good cholesterol, high blood fats and extra fat around the waist. Girls with MBS are at high risk for getting diabetes and heart disease.

DETAILED DESCRIPTION:
Once enrolled in the study, you will have a physical exam done. This includes getting a medical history, height, weight, blood pressure and heart rate. We will also listen to your heart and lungs. We will also look at your skin and determine what stage of puberty you are in by looking at your breast growth and body hair. You will also have two (maybe three) blood tests. The first one is an oral glucose tolerance test (OGTT). During this test, we will have you drink an orange sugary drink and then we will draw your blood. The second test is a frequently sampled intravenous glucose tolerance test (FSIGT). During this test, we will give you insulin through one IV catheter and then we will draw blood from another IV catheter. The third test that you might have done is an ACTH test. During this test, we will draw your blood and then you will be given a dose of cortrosyn (a hormone that your body already makes) and then we will draw your blood again. You will also have two scans of your body done during your visit. There will be a Dual Energy X-Ray Scan (DEXA) and a Magnetic Resonance Imaging Scan (MRI). You will be placed in the machines and then the scanner will move over your body.

ELIGIBILITY:
Inclusion Criteria:

* Relatives with polycystic ovary syndrome
* No relatives with polycystic ovary syndrome
* Overweight
* White non-hispanic girls

Exclusion Criteria:

* Chronic Illness
* Smokers
* Already having periods

Ages: 8 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Overweight girls between the ages of 8 and 12
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2006-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
It is believed that PCOS is inherited. We are trying to look for clinical, blood and/or genetic markers of PCOS in the sisters and daughters of women with PCOS | age 8 until onset of menses

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Dunaif, MD, Principal Investigator — Northwestern University, Chicago, IL
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Urbanek M, Sam S, Legro RS, Dunaif A. Identification of a polycystic ovary syndrome susceptibility variant in fibrillin-3 and association with a metabolic phenotype. J Clin Endocrinol Metab. 2007 Nov;92(11):4191-8. doi: 10.1210/jc.2007-0761. Epub 2007 Sep 4. PMID 17785364